CLINICAL TRIAL: NCT03761732
Title: Islamic Trauma Healing: Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Case Western Reserve University (Other); Seattle Pacific University (Other)
Responsible Party: Principal Investigator, Lori Zoellner, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005522
Record Dates: First submitted 2018-11-14; First posted 2018-12-03 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-02

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This is an active intervention feasibility study, using a pre-post clinical trial design; there is no randomization and no control intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PTSD lay-led group treatment program (Experimental): The group will go through the Islamic Trauma Healing Program
  Interventions: Behavioral: Islamic Trauma Healing

INTERVENTIONS:
Behavioral: Islamic Trauma Healing — 6 session behavioral intervention program designed to reduce PTSD and related symptomatology

SUMMARY:
This study will examine the initial feasibility of a program called Islamic Trauma Healing by conducting a small feasibility study (N = 26) of Islamic Trauma Healing in Somalia on key targets of PTSD, depression, somatic symptoms, and quality of life. The hypothesis is that those in Islamic Trauma Healing will show a reduction of PTSD symptoms, depressive symptoms, and somatic symptoms and show improvement in quality of well-being. Feasibility will also be examined by examining at retention, satisfaction, and community feedback.

DETAILED DESCRIPTION:
Islamic Trauma Healing is a lay-led, small-group intervention specifically targeting healing mental wounds of trauma within mosques. The six-session intervention combines empirically supported exposure-based and cognitive restructuring techniques with Islamic principles. A lay-led, group program promotes community building, acknowledges trauma's impact in the community, and facilitates wider implementation. The program is not referred to as "therapy" or "treatment" for "mental illness." It incorporates community building (e.g., shared tea, supplication), integrated Islamic principles that utilize cognitive restructuring through discussion of prophet narratives (e.g., faith during hard times, Prophet Job [Ayyub]), and exposure therapy through individual prayer, talking to Allah about the trauma. Ultimately, the program will follow a self-sustaining train-the-trainer model, led by group leaders, empowering lay leaders to facilitate healing in their communities. Further, training time is dramatically reduced to two, 4-hour training sessions, focusing on teaching skills of group discussion leading rather than training as a lay therapist or mental health counselor. Preliminary data from a community sample and from initial men's and women's groups show a strong perceived need and match with the Islamic faith, with large effects obtained for pre- to post-group across measures (g = 0.76-3.22). Qualitative analysis identified the intervention as operating on potential mechanisms of connectedness to the community, faith integration, healing, and growth. The preliminary data point to the program being well-received and offering a promising model for delivery of a trauma-focused intervention to Muslim communities. The next steps are examining Islamic Trauma Healing in low and moderate-income Muslim countries, examining the feasibility of implementing this lay-led program.

ELIGIBILITY:
Inclusion Criteria:

* Experienced a DSM-5 trauma at least 12 weeks ago
* Report current re-experiencing or avoidance symptoms
* Islamic faith
* 18-65 year of age

Exclusion Criteria:

* Immediate suicide risk, with intent or plan
* Cannot understand consent/visible cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Zoellner, PhD, Principal Investigator — University of Washington
Locations (2):
- Somalia (2):
  - Borama Mosque, Borama
  - Hargeisa Mosque, Hargeisa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klein AB, Egeh MH, Bowling AR, Holloway A, Ali AA, Abdillahi ZA, Abdi MA, Ibrahim SH, Bootan KH, Ibrahim HI, Ali AM, Tubeec AM, Dolezal ML, Angula DA, Bentley JA, Feeny NC, Zoellner LA. WhatsApp supervision for a lay-led Islamic trauma-focused intervention in Somaliland: Qualitative content analysis. J Trauma Stress. 2023 Feb;36(1):59-70. doi: 10.1002/jts.22882. Epub 2022 Oct 6. PMID 36204779
- [Derived] Zoellner LA, Bentley JA, Feeny NC, Klein AB, Dolezal ML, Angula DA, Egeh MH. Reaching the Unreached: Bridging Islam and Science to Treat the Mental Wounds of War. Front Psychiatry. 2021 Jun 2;12:599293. doi: 10.3389/fpsyt.2021.599293. eCollection 2021. PMID 34149468

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PTSD Lay-led Group Treatment Program
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PTSD Lay-led Group Treatment Program
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 26
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Somalia | 26
PTSD Severity (PDS-5) [Mean (Standard Deviation); unit: score on a scale] | 30.88 (13.76)
Depression Symptoms (PHQ-9) [Mean (Standard Deviation); unit: score on a scale] | 10.42 (4.69)
Somatic Symptoms (SSS-8) [Mean (Standard Deviation); unit: score on a scale] | 8.46 (2.53)
Well-Being (WHO-5) [Mean (Standard Deviation); unit: score on a scale] | 10.00 (6.62)

OUTCOME MEASURES:

1. Primary Outcome: PTSD Scale - Self-Report for DSM-5 (PDS-5; Foa et al., 2016)
Description: PTSD symptoms will be measured using the PTSD Scale - Self-Report for DSM-5 (PDS-5; Foa et al., 2016). Twenty items comprise the PTSD severity scale, with scores ranging from 0 to 80 and higher scores indicating higher PTSD severity. A total score is calculated.
Time Frame: Last 1 Week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PTSD Lay-led Group Treatment Program
Number analyzed (Participants) | 26
score on a scale | 8.08 (5.74)

2. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001)
Description: The PHQ-9 is a self-report measure of depression symptoms with each question rated from 0-3. Higher scores indicate greater depression severity, with scores ranging from 0 to 27.
Time Frame: Last 1 Week
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | PTSD Lay-led Group Treatment Program
Number analyzed (Participants) | 26
score on scale | 2.50 (1.50)

3. Secondary Outcome: Somatic Symptoms Scale-8 (SSS-8; Gierk et al., 2014)
Description: The Somatic Symptoms Scale is an 8 item version of the PHQ-15; self-report assessment of somatic symptoms (e.g., stomach pain, headaches, dizziness). The current version scored items on the original PHQ-15 scale from 0 to 2, with a range from 0 to 16.
Time Frame: Last 1 Week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PTSD Lay-led Group Treatment Program
Number analyzed (Participants) | 26
score on a scale | 2.38 (1.58)

4. Secondary Outcome: Quality of Well-being Index
Description: The WHO-5 Wellbeing Index (WHO-5; Bech, Olsen, Kjoller, & Rasmussen, 2003) will be used to measure well-being. This five-item measure assesses emotional well-being on a 0-5 scale, with higher scores reflecting better well-being. Range of scores is from 0 to 25.
Time Frame: Last 1 Week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PTSD Lay-led Group Treatment Program
Number analyzed (Participants) | 26
score on a scale | 19.38 (2.48)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | PTSD Lay-led Group Treatment Program
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT03761732/Prot_SAP_000.pdf